CLINICAL TRIAL: NCT01887405
Title: Comparative Evaluation of Handling Characteristics of Two Adrenaline Autoinjectors,EpiPen in Comparison With Jext; the HEJ-study
Brief Title: Comparative Evaluation of Handling Characteristics of Two Adrenaline Autoinjectors,EpiPen in Comparison With Jext
Acronym: HEJ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ALK Nordic A/S, Danmark Filial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: JX-A-01
Record Dates: First submitted 2013-06-20; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Handling of Auto-injectors
Keywords: Adrenaline; Auto-injector; Jext; Epipen
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adrenaline: Session 1 Jext, 2 Epipen (Active Comparator): Subjects will be randomised 1:1 to use Jext in session 1 and EpiPen in session 2.
  Interventions: Drug: Adrenaline auto-injector
- Adrenaline: Session 1 Epipen, 2 Jext (Active Comparator): Subjects will be randomised 1:1 to use EpiPen in session 1 and Jext in session 2.
  Interventions: Drug: Adrenaline auto-injector

INTERVENTIONS:
Drug: Adrenaline auto-injector — Each subject will be randomly assigned to use either the Jext or EpiPen first. The alternative auto-injector will then be used by the same subject in the second study session.
  Valid for both Jext and Epipen:
  Active ingredients: Adrenaline tartrate Dosage form: Prefilled auto-injector for single use, delivering one intramuscular injection Dose/strength: 150 μg Excipients: Sodium chloride, sodium metabisulphite (E223), hydrochloric acid (for pH adjustment), water
  Other Names: Jext; Epipen

SUMMARY:
The purpose of the study is to demonstrate non-inferiority of Jext compared with EpiPen for the proportion of subjects with a successful self-injection. And to evaluate and compare the handling characteristics of two auto-injectors (Jext and EpiPen).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before entering the study 1
* Prescription of EpiPen or AnaPen for at least 2 months
* Age ≥16 years
* Body weight >50 kg
* Subject willing and able to comply with study protocol

Exclusion Criteria:

* Any of the following concomitant diseases: cardiovascular disease, e.g. arrhythmias or signs of coronary atherosclerosis, heart failure, uncontrolled hypertension, uncontrolled diabetes mellitus, cancer, hyperthyroidism, severe renal impairment
* Known blood-born infection, e.g. hepatitis and/or HIV
* Concomitant treatment with medication which may potentiate the effect of adrenaline, e.g. catechol-O-methyl transferase (COMT) inhibitors, monoamine oxidase (MAO) inhibitors and tricyclic antidepressants
* Pregnancy
* Being immediate family of the investigator or study staff, defined as the investigator's/staff's spouse, parent, child, grandparent or grandchild

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of Jext compared with EpiPen for the proportion of subjects with a successful self-injection. | 1 day
  The following steps were recorded as correctly done or not by the observer in a check list approach (yes/no):
  1. The subject identified the safety cap.
  2. The subject removed the safety cap.
  3. The subject identified the end of the auto-injector where the needle presents itself
  4. The subject used sufficient force to actuate the injection.
  5. The subject injected the auto-injector into the anterolateral thigh at a right angle (approximately 90°) to the thigh.
  6. The time spent for the injection of adrenaline was more than 10 seconds, i.e. with the needle in situ.
  If all 6 steps were performed correctly, the injection was considered as successful. These data form the basis for evaluation of the binary primary endpoint (successful injection or not).

SECONDARY OUTCOMES:
To evaluate and compare the handling characteristics of two auto-injectors (Jext and EpiPen) regarding subject preference for one of the two auto-injectors over the other, the time to perform the injection and any hesitance to perform the injection | 1 day
  For evaluation of the secondary endpoints, the observer assessed the following:
  The time used for the actuation of the injection, i.e. the time from starting to read the instructions to having injected the adrenaline as recorded by a stop watch. This time was divided into two parts:
  * The time for reading the information
  * The time used to perform the injection Any hesitation from the subject to actuate the injection on a 4-step scale: None, Minor, Severe or Completely Inhibited (i.e. no injection)
  At the end of the second session the subject was asked the following question: "Which auto-injector do you prefer?" The following responses were possible:
  Jext / EpiPen / I don't have any preference for any of the auto-injectors. The preference is a secondary endpoint.

OTHER OUTCOMES:
Evaluation of instructions and AEs | 1 day
  After the injection the subject evaluated the package of instructions (leaflet as well as the information on the auto-injector) for the following (yes/no):
  Were the instructions concise? Were the instructions comprehensible? Do you have any further questions concerning the instructions or do you see any lack of clarity? These have been assessed as other endpoints.
  Safety assessments included recording of all AEs and serious adverse events (SAEs) were done.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Strand, MD Phd, Principal Investigator — Asthma and Allergy Clinic at St Göran's Hospital, Stockholm, Sweden
Locations (1):
- Asthma and Allergy Clinic at St Göran's Hospital, Stockholm, Sweden